CLINICAL TRIAL: NCT03084913
Title: Comparing Diets for Weight Loss and Improvement in Cancer Biomarkers in Men With Prostate Cancer
Brief Title: Olive Oil v Prostate Cancer Foundation Diet for Treatment of Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Mary Flynn, Research dietitian, Associate professor of Medicine, The Miriam Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2134-14
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: dietary treatment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate Cancer Foundation diet (Active Comparator): Intervention: 8-weeks of a Prostate Cancer Foundation diet
  Interventions: Other: Plant- based, olive oil diet; Other: Prostate Cancer Foundation diet
- plant- based, olive oil diet (Experimental): Intervention: 8 weeks of a plant-based, olive oil diet
  Interventions: Other: Plant- based, olive oil diet; Other: Prostate Cancer Foundation diet

INTERVENTIONS:
Other: Plant- based, olive oil diet — used as part of daily diet, followed for 8 weeks
  Other Names: plant-based, olive oil diet
Other: Prostate Cancer Foundation diet — followed for 8 weeks

SUMMARY:
This study compared a plant-based, olive oil diet to the diet recommended by the Prostate Cancer Foundation for weight loss and improvement in some laboratory biomarkers.

DETAILED DESCRIPTION:
Dietary treatment of overweight/ obese men with prostate cancer has not been well studied. As men with prostate cancer who are overweight/ obese are at an increase risk of recurrence, metastasis and mortality, elucidating a diet that will both improve biomarkers for prostate cancer and lead to long-term weight management could improve survivorship. The primary objective of this proposal is to compare a plant-based, olive oil (PBOO) diet to a conventional diet for weight loss and improvement in metabolic biomarkers (specifically fasting insulin, glucose, and triglycerides) for overweight/ obese men diagnosed with prostate cancer on surveillance or who have had an asymptomatic biochemical failure after primary therapy. The secondary objective is to determine which diet will be more acceptable for long term use. Participants will consume for 8 weeks each a conventional diet for treating prostate cancer and a PBOO diet for weight loss and improvement in biomarkers with random assignment to the diet order. They will choose one of the diets for 6 months of follow-up. Blood samples and body weight will be obtained pre- and post diet and after 6 months of follow-up and compared between the diets. Based on earlier work by colleagues of the PI, it is anticipated that the PBOO diet will result in better weight loss and biomarkers and will be more acceptable for long-term weight management. This protocol has the potential to elucidate a diet that will improve the body weight and survival of men with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer, BMI 25.0 to 40.0 kg/m2

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 30 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
weight loss | 8 weeks

SECONDARY OUTCOMES:
improvement in in fasting blood glucose and insulin | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Flynn, PhD, RD, Principal Investigator — Research Dietitian

IPD SHARING:
Plan to Share IPD: No